CLINICAL TRIAL: NCT05641246
Title: Effect of Topical Diclofenac on Clinical Outcome in Breast Cancer Patients Treated With Capecitabine: A Randomized Controlled Trial.
Brief Title: Effect of Topical Diclofenac on Clinical Outcome in Breast Cancer Patients Treated With Capecitabine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: German University in Cairo (Other)
Collaborators: Cairo University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CPH-2022-10-MHS-2
Record Dates: First submitted 2022-11-09; First posted 2022-12-07 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2024-01

CONDITIONS: Hand and Foot Syndrome
Keywords: Capecitabine; Breast Cancer; Hand and Foot Syndrome; Diclofenac Sodium
MeSH Terms: conditions — Hand-Foot Syndrome; Breast Neoplasms | interventions — Urea; Diclofenac

STUDY DESIGN:
Intervention Model Description: The study consists of 2 Arms, A control arm which will only receive standard of care (CARBAMIDE) and an intervention arm which will receive (CARBAMIDE and VOLTAREN)
Who Masked: Participant
Masking Description: The Principle investigator and the Researcher are aware of the intervention taken for each participant. The participant will be blinded ( Single blinded)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Arm (Active Comparator): * Standard of care Urea-based cream (CARBAMIDE®) will be applied to hands and feet 2-3 times daily for 14 days starting from the first dose and cycle of Capecitabine (XELODA ®).
  * Each Capecitabine (XELODA ®) cycle lasts for 21 days.
  * Capecitabine (XELODA ®) dose :2g/m2 daily divided into 2 doses after breakfast and dinner for 14 days followed by 7 days Capecitabine free.
  * Capecitabine (XELODA ®) dose will be modified according to treatment related side effects (26).
  * This regimen will be repeated at each cycle of Capecitabine (XELODA ®) and lasts for 6 cycles (18 weeks) and preventive measures of Hand-foot syndrome will be applied (Avoid mechanical stress
  Interventions: Drug: (CARBAMIDE®)
- Intervention Arm (Active Comparator): * Standard of care Urea-based cream (CARBAMIDE®) will be applied to hands and feet twice daily for 14 days starting from the first dose and cycle of Capecitabine (XELODA ®).
  * Each Capecitabine (XELODA ®) cycle lasts for 21 days.
  * Capecitabine (XELODA ®) dose: 2g/m2 daily divided into 2 doses after breakfast and dinner for 14 days followed by 7 days Capecitabine free.
  * Capecitabine (XELODA ®) dose will be modified according to treatment related side effects (26).
  * This regimen will be repeated at each cycle of Capecitabine (XELODA ®) and lasts for 6 cycles (18 weeks) and preventive measures of Hand-foot syndrome will be applied (Avoid mechanical stress Plus
  * Topical diclofenac (VOLTAREN®) Emulgel 1% 2-4g (2g = 4 fingertip Units (FTU)) twice daily 2 hours away from Urea-based cream (CARBAMIDE®) for 14 days starting from the first cycle and dose of Capecitabine.
  * This regimen will be repeated at each cycle of Capecitabine (XELODA ®) and lasts for 6 cycles (18 weeks).
  Interventions: Drug: (CARBAMIDE®); Drug: (VOLTAREN®) Emulgel 1%

INTERVENTIONS:
Drug: (CARBAMIDE®) — Urea is used to treat dry/rough skin conditions (such as eczema, psoriasis, corns, callus) and some nail problems (such as ingrown nails). It may also be used to help remove dead tissue in some wounds to help wound healing. Urea is known as a keratolytic. It increases moisture in the skin by softening/dissolving the horny substance (keratin) holding the top layer of skin cells together. This effect helps the dead skin cells fall off and helps the skin keep more water in.
  Other Names: Urea-based cream
Drug: (VOLTAREN®) Emulgel 1% — (VOLTAREN®) Emulgel 1% contain the active ingredient diclofenac which belongs to the NSAIDS.it has analgesic and anti-inflammatory properties and due to its alcohol base it has a cooling effect.
  Other Names: Diclofenac Sodium
  Arms: Intervention Arm

SUMMARY:
The aim of the study is to evaluate the efficacy of using combination of Urea-based cream (CARBAMIDE®) and topical diclofenac (VOLTAREN®) Emulgel 1% for improving the incidence of Hand-foot syndrome in histologically proven breast cancer Egyptian patients receiving single agent chemotherapy Capecitabine (XELODA ®) and Its effect on improving patients' quality of life.

DETAILED DESCRIPTION:
Breast cancer (BC) is the most common cancer in women and the leading cause of death associated with cancer in females worldwide. BC, like most cancers, is a heterogeneous disease with a variety of molecular subtypes. Basal-like, Luminal-A, Luminal-B, HER2-positive/HER2-enriched/HER2-overexpressing BC, and normal-like tumors are the major subclasses identified by genetic profiling. Depending on the size, stage, grade, metastatic behavior, aggressiveness and intrinsic molecular subtyping of the tumor, age, menopausal status, overall health, comorbidities, and preferences of the patient, clinicians now have numerous options for breast cancer treatment. Treatment options include chemotherapy, hormone therapy, immunotherapy, radiotherapy, and surgery. The primary treatment option is usually surgery with the goal of complete resection of the major tumor mass. Surgery may be preceded by systemic neoadjuvant therapies to shrink the tumor in preparation for effective surgery and to maximize breast conservation.

The United States FDA has approved a number of drugs for breast cancer therapy, including Capecitabine (Xeloda). However, these drugs are very pricey and have numerous side effects. Patients frequently report decreased appetite, dehydration, diarrhea, Hand-foot syndrome (HFS), irregular periods, mouth and throat sores, nausea, and vomiting as side effects of Capecitabine. These side effects are difficult for patients who are already weakened by the disease to tolerate. Eventually these also affect the decision for further choice of treatment and impair the quality of life. This necessitates the development of novel drugs for the treatment of breast cancer and This is the role of drug repurposing.

The drug repositioning (aka drug repurposing, drug reprofiling, drug re-tasking, drug redesigning, drug resorting, drug reindication, indication switching, therapeutic switching) can be defined as exploring the new uses for an old clinically approved drug, with reduced risk, time and cost. Methotrexate, Raloxifene and Vinblastine are examples of Drug repurposing in breast cancer.

Hand-foot syndrome (HFS) also Known as palmoplantar erythrodysesthesia, is a common side effect of the fluoropyrimidine chemotherapy drug capecitabine. According to reports, 43 % to 71 %of patients receiving single-agent capecitabine chemotherapy have hand-foot syndrome of any grade.

It is characterized initially by palmoplantar numbness, tingling, or burning pain. These symptoms are usually accompanied by clearly defined erythema with or without edema, cracking, or desquamation. Blistering and ulceration may occur in the advanced stages. HFS may manifest as macular hyperpigmentation rather than erythema in people with darker skin (Fitzpatrick skin types V-VI). Symptoms can range from mildly to severely painful.

The pathogenesis of HFS is unclear, but it is assumed to be different for each drug class HFS causes a variety of toxic skin damage, ranging from non-specific scattered keratinocyte necrosis with basal vacuolar degeneration to full epidermal layer necrosis and (sub)epidermal blistering. In addition to eccrine squamous syringometaplasia, inflammation at the dermo-epidermal junction with papillary dermal edema, blood vessel dilation, and a lymphocytic infiltrate has been reported. The unique physiology of the palms and soles may clarify why the effects of these drugs are concentrated in these areas. The palms and soles are highly vascular, with higher rates of skin cell division than other skin areas, as well as high concentrations of eccrine glands and unique temperature modulation.

Unfortunately, no specific guidelines exist for HFS, and only a few randomized trials demonstrating the benefit of topical treatments are available. The most effective way to manage HFS once it has developed is to modify dose intensity in the form of a dose delay or dose reduction, which will affect patients' treatment outcomes and quality of life such as daily activities like walking or using of hands.

The treatment of choice for symptomatic HFS is determined by the severity of symptoms and their impact on Quality of Life (QoL). Vitamin E, steroids (oral dexamethasone), and analgesics are among the systemic treatment options. Current topical treatments are corticosteroids and emollients such as urea-based creams.

Capecitabine and its metabolites are thought to cause COX-2-mediated inflammation; COX-2 inhibition has been shown to be effective in the prevention of HFS. Topical non-steroidal anti-inflammatory inhibitors (NSAIDs), such as diclofenac, can inhibit COX-2 locally and may have a role in reducing HFS, without systemic side effects. However, no study has been conducted to date evaluating the role of topical COX inhibitors in reducing capecitabine-induced HFS. Hence, this study aimed to evaluate the efficacy and safety of topical diclofenac in reducing capecitabine-induced HFS.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 18 years and above.
2. Females.
3. Histologically proven breast cancer patients receiving Capecitabine (XELODA ®) chemotherapy.
4. life expectancy greater than 18 weeks.

Exclusion Criteria:

1. Hypersensitivity to diclofenac, aspirin or other non-steroidal anti-inflammatory drugs (NSAIDS).
2. History of Urticaria.
3. History of acute rhinitis
4. Asthmatic Patients.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Study is conducted on Breast Cancer patients which the majority are females and Males with Breast Cancer are considered rare
Enrollment: 86 (Actual)
Dates: Start 2022-12-08 (Actual); Primary Completion 2023-11-15 (Actual); Study Completion 2023-12-08 (Actual)

PRIMARY OUTCOMES:
• Incidence of HFS between control arm (Urea-based cream (CARBAMIDE®)) and intervention arm (Combination of Urea-based cream (CARBAMIDE®) and (VOLTAREN®) Emulgel 1%) measured by (CTCAE v 5.0). | One year
  • Incidence of HFS between control arm (Urea-based cream (CARBAMIDE®)) and intervention arm (Combination of Urea-based cream (CARBAMIDE®) and (VOLTAREN®) Emulgel 1%) measured by (Common Terminology Criteria for Adverse Effects CTCAE v 5.0).

CONTACTS AND LOCATIONS:
Locations (1):
- KASR ALAINY Center of Oncology and Nuclear medicine, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Harbeck N, Gnant M. Breast cancer. Lancet. 2017 Mar 18;389(10074):1134-1150. doi: 10.1016/S0140-6736(16)31891-8. Epub 2016 Nov 17. PMID 27865536
- [Background] Perou CM, Sorlie T, Eisen MB, van de Rijn M, Jeffrey SS, Rees CA, Pollack JR, Ross DT, Johnsen H, Akslen LA, Fluge O, Pergamenschikov A, Williams C, Zhu SX, Lonning PE, Borresen-Dale AL, Brown PO, Botstein D. Molecular portraits of human breast tumours. Nature. 2000 Aug 17;406(6797):747-52. doi: 10.1038/35021093. PMID 10963602
- [Background] Torre LA, Siegel RL, Ward EM, Jemal A. Global Cancer Incidence and Mortality Rates and Trends--An Update. Cancer Epidemiol Biomarkers Prev. 2016 Jan;25(1):16-27. doi: 10.1158/1055-9965.EPI-15-0578. Epub 2015 Dec 14. PMID 26667886
- [Background] Leidy J, Khan A, Kandil D. Basal-like breast cancer: update on clinicopathologic, immunohistochemical, and molecular features. Arch Pathol Lab Med. 2014 Jan;138(1):37-43. doi: 10.5858/arpa.2012-0439-RA. PMID 24377810
- [Background] Maughan KL, Lutterbie MA, Ham PS. Treatment of breast cancer. Am Fam Physician. 2010 Jun 1;81(11):1339-46. PMID 20521754
- [Background] Davies C, Pan H, Godwin J, Gray R, Arriagada R, Raina V, Abraham M, Medeiros Alencar VH, Badran A, Bonfill X, Bradbury J, Clarke M, Collins R, Davis SR, Delmestri A, Forbes JF, Haddad P, Hou MF, Inbar M, Khaled H, Kielanowska J, Kwan WH, Mathew BS, Mittra I, Muller B, Nicolucci A, Peralta O, Pernas F, Petruzelka L, Pienkowski T, Radhika R, Rajan B, Rubach MT, Tort S, Urrutia G, Valentini M, Wang Y, Peto R; Adjuvant Tamoxifen: Longer Against Shorter (ATLAS) Collaborative Group. Long-term effects of continuing adjuvant tamoxifen to 10 years versus stopping at 5 years after diagnosis of oestrogen receptor-positive breast cancer: ATLAS, a randomised trial. Lancet. 2013 Mar 9;381(9869):805-16. doi: 10.1016/S0140-6736(12)61963-1. PMID 23219286
- [Background] Aggarwal S, Verma SS, Aggarwal S, Gupta SC. Drug repurposing for breast cancer therapy: Old weapon for new battle. Semin Cancer Biol. 2021 Jan;68:8-20. doi: 10.1016/j.semcancer.2019.09.012. Epub 2019 Sep 21. PMID 31550502
- [Background] Akram M, Siddiqui SA. Breast cancer management: past, present and evolving. Indian J Cancer. 2012 Jul-Sep;49(3):277-82. doi: 10.4103/0019-509X.104486. PMID 23238144
- [Background] Paul SM, Mytelka DS, Dunwiddie CT, Persinger CC, Munos BH, Lindborg SR, Schacht AL. How to improve R&D productivity: the pharmaceutical industry's grand challenge. Nat Rev Drug Discov. 2010 Mar;9(3):203-14. doi: 10.1038/nrd3078. Epub 2010 Feb 19. PMID 20168317
- [Background] Pushpakom S, Iorio F, Eyers PA, Escott KJ, Hopper S, Wells A, Doig A, Guilliams T, Latimer J, McNamee C, Norris A, Sanseau P, Cavalla D, Pirmohamed M. Drug repurposing: progress, challenges and recommendations. Nat Rev Drug Discov. 2019 Jan;18(1):41-58. doi: 10.1038/nrd.2018.168. Epub 2018 Oct 12. PMID 30310233
- [Background] Yap YS, Kwok LL, Syn N, Chay WY, Chia JWK, Tham CK, Wong NS, Lo SK, Dent RA, Tan S, Mok ZY, Koh KX, Toh HC, Koo WH, Loh M, Ng RCH, Choo SP, Soong RCT. Predictors of Hand-Foot Syndrome and Pyridoxine for Prevention of Capecitabine-Induced Hand-Foot Syndrome: A Randomized Clinical Trial. JAMA Oncol. 2017 Nov 1;3(11):1538-1545. doi: 10.1001/jamaoncol.2017.1269. PMID 28715540
- [Background] Saif MW, Elfiky AA. Identifying and treating fluoropyrimidine-associated hand-and-foot syndrome in white and non-white patients. J Support Oncol. 2007 Jul-Aug;5(7):337-43. No abstract available. PMID 17708124
- [Background] Kwakman JJM, Elshot YS, Punt CJA, Koopman M. Management of cytotoxic chemotherapy-induced hand-foot syndrome. Oncol Rev. 2020 May 13;14(1):442. doi: 10.4081/oncol.2020.442. eCollection 2020 Feb 18. PMID 32431787
- [Background] Martschick A, Sehouli J, Patzelt A, Richter H, Jacobi U, Oskay-Ozcelik G, Sterry W, Lademann J. The pathogenetic mechanism of anthracycline-induced palmar-plantar erythrodysesthesia. Anticancer Res. 2009 Jun;29(6):2307-13. PMID 19528496
- [Background] Lou Y, Wang Q, Zheng J, Hu H, Liu L, Hong D, Zeng S. Possible Pathways of Capecitabine-Induced Hand-Foot Syndrome. Chem Res Toxicol. 2016 Oct 17;29(10):1591-1601. doi: 10.1021/acs.chemrestox.6b00215. Epub 2016 Sep 28. PMID 27631426
- [Background] Lin E, Morris JS, Ayers GD. Effect of celecoxib on capecitabine-induced hand-foot syndrome and antitumor activity. Oncology (Williston Park). 2002 Dec;16(12 Suppl No 14):31-7. PMID 12520638
- [Background] Kara IO, Sahin B, Erkisi M. Palmar-plantar erythrodysesthesia due to docetaxel-capecitabine therapy is treated with vitamin E without dose reduction. Breast. 2006 Jun;15(3):414-24. doi: 10.1016/j.breast.2005.07.007. Epub 2005 Sep 26. PMID 16188440
- [Background] Drake RD, Lin WM, King M, Farrar D, Miller DS, Coleman RL. Oral dexamethasone attenuates Doxil-induced palmar-plantar erythrodysesthesias in patients with recurrent gynecologic malignancies. Gynecol Oncol. 2004 Aug;94(2):320-4. doi: 10.1016/j.ygyno.2004.05.027. PMID 15297168
- [Background] Murugan K, Ostwal V, Carvalho MD, D'souza A, Achrekar MS, Govindarajan S, Gupta S. Self-identification and management of hand-foot syndrome (HFS): effect of a structured teaching program on patients receiving capecitabine-based chemotherapy for colon cancer. Support Care Cancer. 2016 Jun;24(6):2575-81. doi: 10.1007/s00520-015-3061-6. Epub 2015 Dec 30. PMID 26715292
- [Background] Zhang RX, Wu XJ, Wan DS, Lu ZH, Kong LH, Pan ZZ, Chen G. Celecoxib can prevent capecitabine-related hand-foot syndrome in stage II and III colorectal cancer patients: result of a single-center, prospective randomized phase III trial. Ann Oncol. 2012 May;23(5):1348-1353. doi: 10.1093/annonc/mdr400. Epub 2011 Sep 22. PMID 21940785
- [Background] Santhosh A, Kumar A, Pramanik R, Gogia A, Prasad CP, Gupta I, Gupta N, Cheung WY, Pandey RM, Sharma A, Batra A. Randomized double-blind, placebo-controlled study of topical diclofenac in the prevention of hand-foot syndrome in patients receiving capecitabine (the D-TORCH study). Trials. 2022 May 19;23(1):420. doi: 10.1186/s13063-022-06353-2. PMID 35590388